CLINICAL TRIAL: NCT06227832
Title: An Open-label Study to Determine the Effect of Oral Doses of KP-001 on Metformin and Midazolam Pharmacokinetics After a Single Oral Administration and to Determine the Effect of Clarithromycin on KP-001 Pharmacokinetics After a Single Oral Administration in Healthy Adult Participants
Brief Title: A Study to Determine the Effect of KP-001 on Metformin and Midazolam Pharmacokinetics and the Effect of Clarithromycin on KP-001 Pharmacokinetics in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KP-001-102
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-03

CONDITIONS: Healthy Adults
Keywords: Phase 1; Drug-drug interaction
MeSH Terms: interventions — Metformin; Midazolam; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- KP-001/Metformin (Experimental)
  Interventions: Drug: KP-001; Drug: Metformin
- KP-001/Midazolam (Experimental)
  Interventions: Drug: KP-001; Drug: Midazolam
- KP-001/Clarithromycin (Experimental)
  Interventions: Drug: KP-001; Drug: Clarithromycin

INTERVENTIONS:
Drug: KP-001 — KP-001
Drug: Metformin — oral dose of 850 mg Metformin
  Arms: KP-001/Metformin
Drug: Midazolam — oral dose of 2 mg Midazolam
  Arms: KP-001/Midazolam
Drug: Clarithromycin — oral doses of 1000 mg Clarithromycin
  Arms: KP-001/Clarithromycin

SUMMARY:
The purpose of this study is to determine the Effects of KP-001 on Metformin (a substrate of MATE1) and Midazolam (a substrate of CYP3A4) Pharmacokinetics and the Effect of Clarithromycin (potent CYP3A4/P-gp Inhibitor) on KP-001 Pharmacokinetics in Healthy Adult Participants. The study will also evaluate the safety and tolerability of KP-001 with and without a single dose or multiple doses of an interaction drug. The study comprises 3 parts. Participants will stay in the Clinical Unit during the study, depending on which part they assigned to. Participants will remain at the clinical site for a 13 day/12 night in-house stay (Part 1), a 14 day/13 night in house stay (Part 2), or a 11 day/10 night in-house stay (Part 3).

ELIGIBILITY:
Inclusion Criteria:

1. Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening Visit procedures.
2. Participants who are male or female, 18-55 years of age, inclusive, at screening.
3. Participant is a continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to Day -1 of Treatment Period 1 and throughout the study, based on participant self-reporting and the result of cotinine test at screening and/or Day -1 of Treatment Period.
4. Participant is medically healthy with no clinically significant abnormal screening results (e.g., medical history, physical examination, laboratory profiles, vital signs, or ECGs), in the opinion of the Investigator or designee. If screening and/or admission results are abnormal, they may be repeated once at screening and/or once at admission to confirm the participant's eligibility.
5. Participant has body weight ≥ 50.0 kg and BMI within the range 18.0 to 30.0 kg/m2 (inclusive) at screening.
6. Participant is a woman of non-childbearing potential who:

   1. Is postmenopausal with amenorrhea for at least 1 year prior to screening and with follicle-stimulating hormone (FSH) of 40 IU/L or higher.

      OR
   2. Has undergone one of the following:

      * bilateral tubal ligation or bilateral salpingectomy
      * hysterectomy
      * bilateral oophorectomy
7. Male participant who is sexually active with female partner(s) of childbearing potential must agree to use both a condom and spermicide from the first dose until 91 days after the last dose of KP-001.
8. Male participant must agree not to donate sperm from the first dose until 91 days after the last dose of KP-001.

Exclusion Criteria:

1. Participant is Japanese, Korean or Chinese descent.
2. Participant is legally, mentally or physically incapacitated or, in the opinion of the Investigator, has significant mental or emotional problems, including psychiatric illness (e.g., depression and/or anxiety) at the time of the Screening Visit, or that could reasonably be expected to develop during the conduct of the study.
3. Participant has a significant history or clinical manifestation of any metabolic, allergic, dermatologic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder as determined by the Investigator or designee.
4. Participant has a history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
5. Participant used any prescription or non-prescription medications (including vitamins, recreational drugs, and dietary or herbal supplements) within 14 days or 5 half-lives (whichever is longer) prior to Day -1 of Treatment Period 1 and until completion of the Follow-up visit unless, in the opinion of the Investigator, may be treatment for an adverse event (AE) or will not interfere with the interpretation of safety.
6. Participant underwent blood donation or transfusion within 56 days prior to Day -1 of Treatment Period 1.
7. Participant has a history or presence of hypersensitivity or idiosyncratic reaction to any components of the KP-001 formulation or any components of formulation used as study intervention during the study.
8. Participant has a history of drug or alcohol abuse [regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor) within one year before the Screening Visit.
9. Participant has a complication of drug allergies or history of drug allergies.
10. Female participant has a positive pregnancy test or is lactating.
11. Participant used any investigational drug in the last 30 days or 5 half-lives (if known), whichever is longer, prior to Day -1 of Treatment Period 1.
12. Participant had any major illness within 30 days before the Screening Visit.
13. Participant had any major surgical procedure within 30 days prior to Day -1 of Treatment Period 1 or any planned surgery during study period.
14. Participant had any laboratory abnormality that, in the judgment of the Investigator, would put the participant at unacceptable risk for participation in the study or may interfere with the assessments included in the study.
15. Participant has abnormal findings on the screening ECG deemed clinically significant by the Investigator or qualified designee.
16. Participant is an employee of the Sponsor or any contract research organization (CRO) involved in the study, the Investigator, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.
17. Participant has consumed alcohol- or caffeine-containing foods and beverages within 72 hours prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study, unless deemed acceptable by the Investigator.
18. Participant has positive urine drug or urine alcohol and positive cotinine test results at Screening or Day -1 of Treatment Period 1.
19. Participant has consumed grapefruit-containing foods and beverages within 7 days prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study.
20. Participant has consumed St. John's wort-containing foods and beverages within 14 days prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study.
21. Participant is unable or unwilling to undergo multiple venipunctures.
22. Participant has a history or presence of liver disease or cholecystectomy within one year prior to screening.
23. Participant has an HbA1c >5.7% at Screening.
24. Participant has positive results at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBcAb), hepatitis B core antibody (HBsAg) or hepatitis C virus (HCV).
25. Participant has a disorder or any condition that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
26. Participant has an estimated creatinine clearance calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula <80 mL/min at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters of metformin in plasma: Area under the concentration-time curve from time 0 extrapolated to infinite time (AUCinf) | 13 days
  To assess the effect of repeated doses of KP-001, an inhibitor of organic cation transporter 2 (OCT2) and multidrug and toxin extrusion protein 1 (MATE-1), on the PK of a single dose of metformin in healthy adult, non-east Asian participants in the United States.
PK parameters of midazolam in plasma: AUCinf | 14 days
  To assess the effect of repeated dose of KP-001, an inducer of CYP3A4, on the PK of a single dose of midazolam in healthy adult, non-east Asian participants in the United States.
PK parameters of KP-001 in plasma: AUCinf | 11 days
  To compare the PK of KP-001 administered alone as a single dose and in combination with clarithromycin, an inhibitor of CYP3A4 and P-gp, in healthy adult, non-east Asian participants in the United States.
PK parameters of metformin in plasma: Maximum observed concentration (Cmax) | 13 days
  To assess the effect of repeated doses of KP-001, an inhibitor of organic cation transporter 2 (OCT2) and multidrug and toxin extrusion protein 1 (MATE-1), on the PK of a single dose of metformin in healthy adult, non-east Asian participants in the United States.
PK parameters of midazolam in plasma: Cmax | 14 days
  To assess the effect of repeated dose of KP-001, an inducer of CYP3A4, on the PK of a single dose of midazolam in healthy adult, non-east Asian participants in the United States.
PK parameters of KP-001 in plasma: Cmax | 11 days
  To compare the PK of KP-001 administered alone as a single dose and in combination with clarithromycin, an inhibitor of CYP3A4 and P-gp, in healthy adult, non-east Asian participants in the United States.

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Early Phase Clinical Unit - Los Angeles, Glendale, California, United States